CLINICAL TRIAL: NCT05359458
Title: The Effect of Emotional Freedom Liberation Technique on Surgical Fear and Anxiety Applied to Patients Before Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Emotional Freedom Liberation Technique, Surgical Fear and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayşegül Yayla, Asistant Professors, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AEP17
Record Dates: First submitted 2022-04-11; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Emotional Distress
Keywords: surgery; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Freedom Liberation Technique Applied to Laparoscopic Cholecystectomy Patients (Experimental): The intervention group is the group in which the investigators applied Emotional Freedom Liberation Technique Intervention: Behavioral: Emotional Freedom Liberation Technique
  Interventions: Behavioral: Emotional Freedom Liberation Technique
- Standard Clinical Care Applied to Laparoscopic Cholecystectomy Patients (No Intervention): The control group is the group that receives standard clinical care

INTERVENTIONS:
Behavioral: Emotional Freedom Liberation Technique — The investigators will apply Emotional Freedom Liberation Technique
  Arms: Emotional Freedom Liberation Technique Applied to Laparoscopic Cholecystectomy Patients

SUMMARY:
Aim: In this study, the effect of Emotional Freedom Technique applied to patients before Laparoscopic Cholecystectomy on surgical fear and anxiety was investigated.

Design: This is a randomized controlled study. Method: A total of 112 patients who were going to have Laparoscopic Cholecystectomy were randomly divided into two groups each including 56 participants. The intervention group was provided with Emotional Freedom Technique. The control group received routine face-to-face education. Surgical fear and anxiety were examined.

ELIGIBILITY:
Inclusion Criteria:

* Clinical treatment for Laparoscopic Cholecystectomy
* 18 years of age or older
* Mentally healthy

Exclusion Criteria:

* Agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Surgical Fear Scale | through study completion, an average of 5 month
  Surgical Fear Scale will be filled in the preoperative period. ll items are scored on an eleven point numeric rating scale (NRS) ranging from 0 (not at all afraid) to 10 (very afraid). This results in a score of 0-40 for each subscale and a total score of 0 to 80.

SECONDARY OUTCOMES:
Anxiety Scale | through study completion, an average of 5 month
  Anxiety scale will be filled in the preoperative period. The scale consists of 10 statements that include the fears that patients may experience about the surgery. The maximum score that can be obtained from the scale is 50. High scores in scale scoring reflect concerns about pain, death during surgery, and postoperative complications and limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, ABD Veya Kanada'da Lütfen Seçin ..., Turkey (Türkiye)